CLINICAL TRIAL: NCT00409500
Title: A Randomized, Double-Blind, Placebo-Controlled, Interleaved, Ascending Dose Study, to Evaluate Safety, Tolerability and Pharmacokinetics of Single Oral Doses of AQW051; to Evaluate the Effect of Food on the Pharmacokinetics of AQW051, in Japanese Healthy Male Subjects
Brief Title: Effect of Food on the Pharmacokinetics of AQW051 in Japanese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAQW051A1101
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: Safety, tolerability, pharmacokinetics, AQW051, food, Japanese, healthy male subjects; Healthy volunteers study
MeSH Terms: interventions — 3-(6-p-tolylpyridin-3-yloxy)-1-azabicyclo(2.2.2)octane

INTERVENTIONS:
Drug: AQW051

SUMMARY:
This study will evaluate safety, tolerability and pharmacokinetics of individual oral doses of AQW051 in Japanese healthy male subjects, and will also evaluate the effect of food on the pharmacokinetics of AQW051.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy male subjects age 20 to 45 years of age, and in good health
* At screening and baseline, the subjects must be in good health as determined by past medical history, physical examination, electrocardiogram, laboratory tests and urinalysis.
* Body mass index within the range of 17 to 25 kg/m2 and weigh at least 50 kg

Exclusion Criteria:

* Smokers (use of tobacco products in the previous 3 months). Urine cotinine levels will be measured during screening for all subjects. Smokers will be defined as any subject who reports tobacco use or has a urine cotinine 'high' level in checking by NicCheck® I.
* Use of any prescription drugs within 4 weeks prior dosing, or over-the-counter medication (vitamins, herbal supplements, dietary supplements) within 2 weeks prior to dosing. Acetaminophen is acceptable.
* Participation in any clinical investigation within 4 months prior to study start.
* Donation or loss of 400 mL or more of blood within 3 months; donation or loss of 200 mL or more of blood within 1 month; or donation of component blood within 2 weeks prior to study start.
* Subjects considered unsuitable for participation in the study within 2 weeks prior to dosing.
* A past medical history of clinically significant abnormality detected during electrocardiogram (ECG) examination or an evident family history (grandparents, parents and siblings) of a ECG abnormality (i.e. prolonged QT-interval syndrome).
* History of fainting, hypotension when standing up, arrhythmia.
* History of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
* History of clinically significant drug allergy, history or presence of atopic allergy (asthma, urticaria, eczematous dermatitis) unless inactive seasonal allergy, or history of food allergy. A known hypersensitivity to the study drug or drugs similar to the study drug.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject in case of participation in the study.
* History of immunodeficiency diseases, including a positive HIV test result.
* A positive Hepatitis B surface antigen (HBsAg), Hepatitis C or Syphilis test result.
* History of drug or alcohol abuse within the 12 months prior to study participation or evidence of such abuse as indicated by the laboratory assays conducted at screening.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54
Dates: Start 2006-10

PRIMARY OUTCOMES:
Safety and tolerability of single oral doses of AQW051 in Japanese healthy male subjects at the end of the study

SECONDARY OUTCOMES:
Pharmacokinetics of single oral doses of AQW051 in Japanese healthy male subjects at the end of the study
Effect of food on the pharmacokinetics of AQW051 after each dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Japan, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Tokyo, Japan